CLINICAL TRIAL: NCT05468541
Title: Psychological and Quality of Life Impact of Brain in Hand
Acronym: BraininHand
Status: Completed | Type: Observational
Sponsor: Cornwall Partnership NHS Foundation Trust (Network)
Collaborators: braininhand.co.uk (Unknown)
Responsible Party: Sponsor
Other Study IDs: Version 4 25.10.21
Record Dates: First submitted 2022-06-22; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective cohort mixed study using both qualitative and quantitative elements. The quantitative component will involve tracking outcomes at baseline and at twelve weeks, using Health of the Nation Outcome Scale for People with a Learning Disability (for quality of life) and Hospital Anxiety and Depression Rating Scale (for anxiety and depression). The qualitative study will involve semi structured interviews with end users to understand usage and acceptability of Brain in Hand app with the added impact of the pandemic.

DETAILED DESCRIPTION:
The Brain in Hand App (BiH) has been awarded a Small Business Research Initiatives competitive grant to develop and test new technologies for the NHS https://braininhand.co.uk/news/brain-in-hand-wins-sbri-healthcare-award/ .

A cohort study is needed to robustly test the BiH technology to evaluate the influence, understand its capabilities, users' experiences, and the effect of clinical impact by looking to align or use the NICE Evidence Framework for Health Digital Technologies, to reference the strengths, weakness, and limitations of BiH specifically around psychological wellbeing and by extension, quality of life. This is the purpose of the study.

There are more than 700,000 autistic people in the United Kingdom. Autism research has focused on causes of autism and largely missed opportunities to discover what helps autistic people. Research highlights that autistic people experience poor mental and physical health, which go unrecognised. Autistic people have very high rates of comorbid physical disabilities as well as mental health conditions that are impacted bilaterally by the social environment. ASD is unique to the person, so person centred support is needed, and a digital solution may offer the best solution in terms of privacy and cost.

NHS England recently reported autistic people have high levels of unmet needs and existing health and social services do not usually cater for this complex group, to deliver person centred support. BiH has developed remote person-centred support with self-management tools with 24/7 helpline that encompasses a wraparound healthcare service. This has recently acquired a further interesting dimension as remote interventions have facilitated enhanced accessibility to healthcare during the pandemic.

The study participants will complete two questionnaires: The self-reporting Hospital Anxiety and Depression Scale and the quality of life, Health of the Nation Scale for people with Learning Disabilities. The questionnaires will gather baseline data and then three months later the same questionnaires will be repeated to understand change. Semi-structured questions will be utilised on a randomly selected sample from the main cohort to gain a user's experience of clinical need and safety.

ELIGIBILITY:
Inclusion Criteria:

1. All who have been diagnosed with Autism Spectrum Disorder (ASD) as per DSM-5 criteria level (1) or post screening by health professional such as a GP and on the confirmatory diagnostic pathway.
2. Age ranges from 19 to 80.
3. Participant has been screened by the Columbia Suicide Rating Scale as not having risk concerns of suicide.
4. Access to smart devices with compatibility to running BiH. The Participant will require a Smart Phone and either a Laptop / Tablet / Note Book.
5. Has capacity to give informed consent and can give informed consent.
6. They can understand the BiH information.

Exclusion Criteria:

1. Outside of stated age range within the inclusion criteria.
2. Any acute or chronic condition, particularly neurodevelopmental conditions such as significant intellectual disability, Level 2/3 DSM V ASD.
3. Diagnosed con-current psychological comorbidity (psychosis, severe depression etc.) that would limit the ability of the participant to take part in the study.
4. Anyone who declines to give consent or are unable to give informed consent. 5. Anyone who has been screened positive with the (C-SSRS) suicide risk scale.

6. Not willing to engage with smart device/internet. 7. Insufficient English language to understand and complete questionnaires.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the participant's existing clinical care team will access their patient records and their autism waiting list to identify potential participants for the study with the participation criteria followed without deviation.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
What is the impact of BiH on quality of life over a three-month period? | 3 months
  The Health of the Nation Outcome Scales for People with Learning Disabilities is measured on a five-point scale (0-4) with 0 being no problem and 4 being very severe. It is completed at Baseline and 3 months and the scores will be compared
What is the impact of BiH on the participant's mental health? | 3 months
  Hospital Anxiety and Depression Scale is measured on a four-point scale (0-3) with 0 being no problem and 4 being very severe. It is completed at Baseline and 3 months and the scores will be compared
Level of acceptability (drop-out rates) | 3 months
  Drop out rates will be recorded
Discover the participant's experience of using BiH App to measure outcomes of reliance on their care support | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
Understand how BiH impacts on coping skills | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
To gain understanding of how BIH has impacted on the autistic person's ability to manage challenging social situations | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
Does BiH App help autistic people feel safe? | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
Does the BiH help autistic people feel more independent? | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
Can access 24/7 telephone support help autistic people feel self-empowered to manage their anxiety? | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
To gain an understanding of how BiH Traffic Light system helps a person manage their anxiety, independence and support their coping skills | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability
Does the participant believe remote support has improved their access to healthcare during the pandemic? | 3 months
  Short semi structured interviews with ten end users to understand usage and acceptability

CONTACTS AND LOCATIONS:
Locations (1):
- Cornwall Partnership NHS Foundation Trust, Bodmin, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No